CLINICAL TRIAL: NCT03629990
Title: Approach Bias Modification for the Treatment of Cannabis Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00077532; 5K23DA045099-05 (NIH)
Record Dates: First submitted 2018-05-16; First posted 2018-08-14 (Actual); Results first posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Cannabis Use Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active ABM + CBT/MET (Experimental): Participants in the Active ABM condition will receive approach bias modification (ABM) training sessions aimed at reducing cognitive bias for cannabis cues.
  All participants will receive MET/CBT therapy.
  Interventions: Behavioral: Approach Bias Modification (ABM); Behavioral: Psychosocial therapy for cannabis use disorder.
- Sham ABM + CBT/MET (Sham Comparator): Participants in the Sham ABM condition will undergo similar computerized tasks without the manipulation of response contingencies that target modification of approach bias.
  All participants will receive MET/CBT therapy.
  Interventions: Behavioral: Sham ABM; Behavioral: Psychosocial therapy for cannabis use disorder.

INTERVENTIONS:
Behavioral: Approach Bias Modification (ABM) — Approach bias modification (ABM) is a novel treatment that involves retraining the implicit action tendency to approach a drug cue by manipulating contingencies in a stimulus-response paradigm.
  Arms: Active ABM + CBT/MET
Behavioral: Sham ABM — Sham ABM involves similar computerized procedures that mimic the active experimental condition, but do not involve manipulation of response contingencies and thus it does not contain any "active" intervention.
  Arms: Sham ABM + CBT/MET
Behavioral: Psychosocial therapy for cannabis use disorder. — All participants will receive psychosocial therapy for cannabis use disorder.

SUMMARY:
Effective and durable treatments for cannabis use disorder remain elusive. Given the increasing prevalence rates of cannabis use and CUD nationwide, investigation of novel treatments is warranted. Implicit cognitive processing is an emerging, and potentially critical therapeutic target.

Cognitive models of addiction posit an override of explicit control-related cognitive processes by implicit reward-driven processes resulting from chronic drug exposure. One form of implicit cognitive processing is approach bias, or, the automatic tendency to approach rather than avoid drug cues, which has been identified for alcohol, nicotine, opioids, and cannabis. Cannabis approach bias predicts increased cannabis use, dependence severity, and cannabis-related problems among heavy cannabis users. Approach bias modification (ABM) is a novel treatment approach that seeks to reduce approach bias by attenuating the incentive-salience of drug cues, and subsequently, drug cue reactivity and drug use. ABM has been shown to reduce relapse rates in alcohol dependent adults by 10-13% at one-year follow-up, and dependence severity in nicotine dependent adults. Our pilot data suggests that ABM may also reduce cannabis craving and that gender may moderate the effect of ABM on cannabis sessions per day in non-treatment seeking adults with CUD. A recent fMRI study with alcohol-dependent adults found decreased mesolimbic activation in participants who received ABM compared to sham-control participants. ABM appears to target implicit reward-driven processes, and could be an effective adjunct to traditional psychosocial and/or future pharmacological interventions that target explicit control-related processes.

Building on our promising feasibility data, the proposed K23 research study will examine the effects of ABM on cue-reactivity and cannabis outcomes in a four-session randomized, double-blind, sham-controlled pilot treatment trial. One-hundred and six (106) treatment-seeking adults with moderate to severe CUD will be randomized to receive either MET/CBT plus ABM or Motivational Enhancement Therapy/Cognitive Behavioral Therapy(MET/CBT) plus sham-ABM. An equal number of men and women will be recruited and randomization will be stratified by gender. ABM sessions will occur following each of the three weekly MET/CBT therapy sessions. Primary outcomes will include cannabis cue-reactivity and cannabis use.

ELIGIBILITY:
Inclusion Criteria:

1. Be age 18-65 and must be able to provide informed consent.
2. Meet DSM-5 criteria for current moderate to severe CUD (past 60 days).
3. Identify cannabis as their primary substance of choice.
4. Consent to remain abstinent from alcohol and cannabis for 12 hours immediately prior to study visits and other drugs of abuse (except nicotine) for three days prior (see Additional Instrumentation below for methods); by restricting cannabis and other substance use as proposed, participants should not be under the acute effects of cannabis or other substances.

Exclusion Criteria:

1. Evidence of, or a history of serious medical or neurological disease that may affect cognitive processing.
2. History of, or current psychotic disorder, bipolar disorder, and attention-deficit hyperactivity disorder, or current untreated major depressive disorder as these may interfere with subjective measurements.
3. Current use of psychotropic medications because these may affect subjective measurements (individuals taking antidepressants will be allowed).
4. Current suicidal ideation. Individuals who endorse suicidal ideation will be seen by a psychologist or psychiatrist in the office and will be referred to treatment as necessary.
5. Women who are pregnant, nursing or of childbearing potential and not practicing an effective means of birth control.
6. Moderate to severe DSM-5 substance use disorder within the past 60 days (other than nicotine or cannabis).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Sherman, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medial University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Active ABM + CBT/MET: Participants in the Active ABM condition will receive approach bias modification (ABM) training sessions aimed at reducing cognitive bias for cannabis cues.
  All participants will receive MET/CBT therapy.
  Approach Bias Modification (ABM): Approach bias modification (ABM) is a novel treatment that involves retraining the implicit action tendency to approach a drug cue by manipulating contingencies in a stimulus-response paradigm.
  Psychosocial therapy for cannabis use disorder.: All participants will receive psychosocial therapy for cannabis use disorder.
- Sham ABM + CBT/MET: Participants in the Sham ABM condition will undergo similar computerized tasks without the manipulation of response contingencies that target modification of approach bias.
  All participants will receive MET/CBT therapy.
  Sham ABM: Sham ABM involves similar computerized procedures that mimic the active experimental condition, but do not involve manipulation of response contingencies and thus it does not contain any "active" intervention.
  Psychosocial therapy for cannabis use disorder.: All participants will receive psychosocial therapy for cannabis use disorder.
Period: Overall Study
Arm/Group | Active ABM + CBT/MET | Sham ABM + CBT/MET
Started | 53 | 51
Completed | 26 | 29
Not Completed | 27 | 22

BASELINE CHARACTERISTICS:
Population: Baseline analysis population consists of all participants successfully randomized either active or sham condition.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active ABM + CBT/MET | Sham ABM + CBT/MET | Total
Number analyzed (Participants) | 53 | 51 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 52 | 50 | 102
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (11.7) | 31.1 (10) | 32.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 29 | 28 | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 15 | 28
  White | 37 | 33 | 70
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 53 | 51 | 104
Marijuana Craving Questionnaire Total Score (MCQ) [Mean (Standard Deviation); unit: units on a scale] — Cannabis craving was assessed using the Marijuana Craving Questionnaire-Short Form (MCQ-SF) a self-reporting tool with 12 items rated on a 7-point Likert scale from 1 (strongly disagree) to 7 (strongly agree). The 12 items are grouped by certain characteristics and the score of each of resulting groups correlates to the intensity of the four craving dimensions (compulsivity, emotionality, expectancy, and purposefulness). Scores from the four subscales are summed with total possible scores ranging from 12 - 84. Higher scores are indicative of increased craving. Population: Baseline analysis on n=98 participants that returned to have MCQ assessment on visit 1. Data are presented as baseline measures on visit 1.
  units on a scale
    number analyzed (Participants) | 50 | 48 | 98
    (all) | 42.5 (16.0) | 41.9 (14.5) | 42.2 (15.2)

OUTCOME MEASURES:

1. Primary Outcome: Cannabis Approach Bias
Description: Using a cue-reactivity paradigm, we will evaluate the efficacy of approach bias modification on cannabis approach bias.
  Participants are presented with cannabis related and neutral images on a computer screen and are asked to push or pull a joystick in response to a non-content related stimulus feature (i.e. image border color - blue or yellow). Joystick movement activates a zooming feature, which has been shown to effectively simulate approach (pull-zoom in) and avoidance (push-zoom out), and reaction times are calculated from image onset to zoom off-screen. Participants are asked to respond as quickly and accurately as possible. Cannabis approach bias is computed by subtracting "pull CB cue" reaction times (RTs) from "push CB cue" RTs (CBpushRT - CBpullRT); a positive value thus indicates greater cannabis approach bias. Approach bias assessments occurred at 3 time points: baseline (pre-assessment), end of study (post-assessment), and follow-up (follow-up assessment). During t
Time Frame: Baseline, End of Treatment (4 weeks), Follow-Up (8 weeks)
Population: All randomized participants with at least one post randomization visit.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active ABM + CBT/MET | Sham ABM + CBT/MET
Number analyzed (Participants) | 50 | 48
seconds
  Baseline: neutral | -8.43 (57.1) | 4.05 (46.1)
  Baseline: cannabis | 5.43 (56.2) | -1.36 (41.9)
  End of Treatment (4 weeks): neutral: number analyzed (Participants) | 35 | 37
  End of Treatment (4 weeks): neutral | 1.8 (43.6) | -0.22 (49.3)
  End of Treatment (4 weeks): cannabis: number analyzed (Participants) | 35 | 37
  End of Treatment (4 weeks): cannabis | -16.1 (41.9) | -1.74 (47.8)
  Follow Up (8 weeks): Neutral: number analyzed (Participants) | 25 | 29
  Follow Up (8 weeks): Neutral | 2.82 (47.8) | -6.34 (33.7)
  Follow Up (8 weeks): Cannabis: number analyzed (Participants) | 25 | 29
  Follow Up (8 weeks): Cannabis | -6.76 (29.4) | 1.66 (24.3)

2. Secondary Outcome: Percent Days Using Cannabis
Description: Using self-report we will evaluate the efficacy of ABM on percent days using cannabis, measurements will be summarized at end of study treatment and at the follow up visit.
Time Frame: Baseline, End of Treatment (4 weeks), Follow-Up (8 weeks)
Population: all randomized participants that returned post randomization.
Measure: Mean (Standard Deviation); unit: Percentage of day reported using can
Arm/Group | Active ABM + CBT/MET | Sham ABM + CBT/MET
Number analyzed (Participants) | 50 | 48
Percentage of day reported using can
  Baseline | 86.6 (20.2) | 87.7 (18.9)
  End of Treatment (4 weeks): number analyzed (Participants) | 36 | 37
  End of Treatment (4 weeks) | 74.1 (29.1) | 72.0 (28.4)
  Follow Up (8 weeks): number analyzed (Participants) | 25 | 29
  Follow Up (8 weeks) | 69.1 (35.3) | 71.7 (34.8)

3. Secondary Outcome: Marijuana Craving Questionnaire Total Score (Craving)
Description: Cannabis craving was assessed using the Marijuana Craving Questionnaire-Short Form (MCQ-SF) a self-reporting tool with 12 items rated on a 7-point Likert scale from 1 (strongly disagree) to 7 (strongly agree). The 12 items are grouped by certain characteristics and the score of each of resulting groups correlates to the intensity of the four craving dimensions (compulsivity, emotionality, expectancy, and purposefulness). Scores from the four subscales are summed with total possible scores ranging from 12 - 84. Higher scores are indicative of increased craving.
Time Frame: 8 weeks
Population: All randomized participants that have at least 1 time point of MCQ measured.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active ABM + CBT/MET | Sham ABM + CBT/MET
Number analyzed (Participants) | 50 | 48
units on a scale
  Baseline: Non MJ | 39.5 (16.1) | 38.6 (16.2)
  Baseline: MJ | 43.1 (17.8) | 40.3 (17.6)
  End of Treatment (4 weeks): Non MJ: number analyzed (Participants) | 36 | 35
  End of Treatment (4 weeks): Non MJ | 31 (15.9) | 31.1 (15.8)
  End of Treatment (4 weeks): MJ: number analyzed (Participants) | 36 | 35
  End of Treatment (4 weeks): MJ | 31.4 (13.9) | 32.1 (17.2)
  Follow up (8 weeks): Non MJ: number analyzed (Participants) | 25 | 29
  Follow up (8 weeks): Non MJ | 28.3 (16.9) | 25.2 (14.5)
  Follow Up (8 weeks): MJ: number analyzed (Participants) | 25 | 29
  Follow Up (8 weeks): MJ | 30 (18.5) | 26.5 (15.1)

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Active ABM + CBT/MET | Sham ABM + CBT/MET
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/51
Other Adverse Events (participants affected / at risk) | 0/53 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT03629990/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT03629990/ICF_001.pdf